CLINICAL TRIAL: NCT06277817
Title: The Effect of Chest Physiotherapy Techniques Applied Before Aspiration on Vital Signs, Blood Gas Values and Secretion Amount in Patients on Mechanical Ventilation Support
Brief Title: The Effect of Chest Physiotherapy Methods Applied Before Aspiration on Respiratory Characteristics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Serap Parlar Kılıç, Proffessor, Inonu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2021/1916
Record Dates: First submitted 2023-04-02; First posted 2024-02-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Patient Involvement
Keywords: Expiratory rib cage compressio; Chest physiotherapy; Mechanical ventilation; Percussion-Vibration; Intensive care
MeSH Terms: conditions — Patient Participation

STUDY DESIGN:
Intervention Model Description: The randomization of this study was performed by a statistical expert independent of the study, using the computer-assisted Random Allocation Rule method, which is one of the random assignment methods (http://biostatapps.inonu.edu.tr/RAY/).78 patients to be included in the study were divided into 3 groups and assigned an equal number of patients in each group according to the results of the random assignment method. In order to assign patients to research groups impartially, the research groups determined were written on papers and group assignments were made by drawing lots. Thus, the number of individuals in the groups and the probability of each patient included in the study being in either of the experimental or control groups were equalized.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- expiratory rib cage compression group (Experimental): Expiratory rib cage compression procedure phase; Three hours after the first aspiration data were obtained, before the second aspiration, expiratory rib cage compression was applied for 5 minutes in the right lateral and left lateral positions, applying to both lungs, with the most affected lung area first. Before and after the procedure, vital signs, blood gas parameters were measured and the amount of secretion collected during the aspiration process was weighed.
  Interventions: Other: expiratory rib cage compression
- percussion vibration group (Experimental): Percussion, vibration process stage; Three hours after the first aspiration data were obtained, before the second aspiration, percussion and vibration were applied 3-5 times to each area, starting from the right and left lower lobes, in the right lateral and left lateral positions, with the most affected lung area being applied to both lungs first. Vital signs, blood gas parameters were measured before and after the procedure, and the amount of secretion collected during the aspiration process was weighed.
  Interventions: Other: percussion vibration
- control group (No Intervention): Control group phase; In this group, vital signs, blood gases, and secretion amount were recorded at the same time as the experimental groups, without any intervention.

INTERVENTIONS:
Other: expiratory rib cage compression — Expiratory rib cage compression: The hands are placed on the lower third of the rib cage. During expiration, the end and sides of the patients' rib cage are gradually compressed with the hands.At the end of expiration, compression is released from the thorax to allow patients to take a free inspiration. After each compression, the patient is allowed to perform 3 breathing cycles.Expiratory rib cage compression is applied for 5 minutes.
  Arms: expiratory rib cage compression group
Other: percussion vibration — Percussion :Percussion is performed 3-5 times on each area from a height of approximately 10 cm with the domed hand. . It starts from the right and left lower lobes and goes up.Vibration:The hand is firmly/strongly placed on the application area. The arm and shoulder are stretched and the fingers are gently vibrated or shaken gently. While the patient is exhaling, vibration is performed 3-5 times in each area, starting from the right and left lower lobes.
  Arms: percussion vibration group

SUMMARY:
Physiotherapy is one of the most frequently used supportive treatments in intensive care units due to its positive effects on critically ill patients. Chest physiotherapy (GF), which constitutes the most effective part of the physiotherapy programs applied to intensive care patients under mechanical ventilation (MV) support, consists of a series of techniques aimed at clearing airway secretions, facilitating appropriate lung ventilation by increasing lung volume and respiratory muscle strength, and improving the respiratory system and gas exchange. . Of these techniques, manually applied percussion vibration and expiratory rib cage compression (EGCC) are some of the most commonly applied GF techniques in patients on MV support. This study was conducted to evaluate the effect of chest physiotherapy techniques applied before aspiration on vital signs, blood gas values and amount of secretion in patients on mechanical ventilation support.

DETAILED DESCRIPTION:
This study was carried out to determine the effect of chest physiotherapy techniques applied before aspiration on the vital signs, blood gas values and amount of secretion in patients on mechanical ventilation support.This randomized, controlled and experimental study was conducted between May 2021 and October 2022 in Tunceli State Hospital intensive care units with patients on mechanical ventilation support. The study was completed with a total of 78 patients, including the percussion vibration group (n=26), the expiratory rib cage compression group (n=26), and the control group (n=26). Data were collected with the "Patient Identification Form", "Vital Signs Recording Form", "Blood Gas Values Recording Form" and "Secretion Amount Recording Form". Two aspirations were performed in each of the three groups with an interval of three hours. Three hours after the first aspiration, chest physiotherapy techniques were applied to the two experimental groups, but not to the control group. A second aspiration was then performed. Vital signs and blood gases were measured before and after both aspiration procedures, and the amount of secretion collected during the two aspiration procedures was weighed.In the comparison between groups according to time; Statistically significant changes were found in heart rate during the first aspiration period, and diastolic blood pressure and respiratory rate during the second aspiration period (p<0.05). In the independent comparison between groups; statistically significant difference was found in diastolic blood pressure, respiratory rate and peripheral SpO2 values (p<0.05). In group comparisons; while the averages of secretion weight and amount did not show a significant change in all three groups (p>0.05), it was found that it tended to increase in the percussion-vibration and expiratory rib cage compression groups, while it tended to decrease in the control group.In this study, it was concluded that chest physiotherapy techniques had a beneficial effect on some vital signs in patients on mechanical ventilation support, did not make any difference in other parameters. Further studies are needed to determine the positive effects of these techniques on vital signs, blood gases and secretion.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Intubated in the intensive care unit for more than 48 hours
* Followed in synchronized intermittent mechanical ventilation (SIMV) mode
* with arterial catheter
* with hemodynamic stability
* PEEP <10
* Patients with Glasgow Coma Scale >3 were included.

Exclusion Criteria:

* Rib fracture, chest trauma
* with pneumothorax
* with hemoptysis
* with increased intracranial pressure
* Having a history of spine surgery
* with chest drainage tube
* Those with skin infection and subcutaneous emphysema in the back and chest area
* The mechanical ventilation setting to be changed during the study
* with life-threatening cardiac arrhythmia
* pregnant
* Obese (Body Mass Index >30)
* Patients who had to be aspirated outside of the specified periods during the study were excluded from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2021-05-19 (Actual); Primary Completion 2021-06-25 (Actual); Study Completion 2022-10-24 (Actual)

PRIMARY OUTCOMES:
The effect of percussion vibration on the amount of secretion | about a year
  Pecussion vibration was applied before endotracheal aspiration, and the secretion accumulated in the collection container during the aspiration process was weighed and recorded.
Effect of expiratory rib cage compression on the amount of secretion | about a year
  Expiratory rib cage compression was applied before endotracheal aspiration, and the secretion accumulated in the collection container during the aspiration process was weighed and recorded.
Effect of percussion vibration on blood gas parameters | about a year
  Percussion vibration was applied before endotracheal aspiration. Measurements of pO2, pH, pCO2, HCO3, SaO2 parameters were recorded 5 minutes before endotracheal aspiration and 25 minutes after applying percussion vibration
Effect of expiratory rib cage compression on blood gas parameters | about a year
  Expiratory rib cage compression was applied before endotracheal aspiration. Measurements of pO2, pH, pCO2, HCO3, SaO2 parameters were recorded 5 minutes before endotracheal aspiration and 25 minutes after applying expiratory rib cage compression.
Perküsyon vibrasyonun yaşam bulgularına etkisi | about a year
  Percussion vibration was applied before endotracheal aspiration. Vital signs measurements of systolic blood pressure, diastolic blood pressure, respiratory rate, pulse rate, body temperature, and peripheral SpO2 were recorded 5 minutes before endotracheal aspiration and 15 minutes after applying percussion vibration.
Effect of expiratory rib cage compression on vital signs | about a year
  Expiratory rib cage compression was applied before endotracheal aspiration. Vital signs measurements such as systolic blood pressure, diastolic blood pressure, respiratory rate, pulse rate, body temperature, and peripheral SpO2 were recorded 5 minutes before endotracheal aspiration and 15 minutes after applying expiratory rib cage compression.

CONTACTS AND LOCATIONS:
Locations (1):
- Tunceli State Hospital, Tunceli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Derived] Olmaz D, Parlar Kilic S. Effects of Pre-Aspiration Chest Physiotherapy Techniques on Vital Signs, Blood Gas Values and Secretions in Mechanically Ventilated Patients. Nurs Crit Care. 2026 Jan;31(1):e70232. doi: 10.1111/nicc.70232. PMID 41536156